CLINICAL TRIAL: NCT02785263
Title: Patient Centered Radiation Treatment of Anal Cancer Using Shared Decision Making as to Dose Level
Brief Title: Shared Decision Making With Anal Cancer Patients on Radiation Dose
Acronym: PC-Anal-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PC-Anal-01
Record Dates: First submitted 2016-05-09; First posted 2016-05-27 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Anal Cancer
Keywords: Anal cancer; Shared decision making
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard radiotherapy (Other): Daily on weekdays: 2.15 gray for tumor and verified lymph node metastases and 1.8 gray for the elective volume. A total of 28 treatments
  Interventions: Radiation: 2.15 gray and 1.8 gray. Max. 6 weeks.
- High dose radiotherapy (Other): Daily on weekdays: 2.15 gray for tumor and verified lymph node metastases and 1.8 gray for the elective volume. A total of 28 treatments
  Interventions: Radiation: 2.15 gray and 1.8 gray. Max. 6 weeks.
- Low dose radiotherapy (Other): Daily on weekdays: 2.15 gray for tumor and verified lymph node metastases and 1.8 gray for the elective volume. A total of 25 treatments
  Interventions: Radiation: 2.15 gray and 1.8 gray. Max. 5 weeks.

INTERVENTIONS:
Radiation: 2.15 gray and 1.8 gray. Max. 6 weeks.
  Arms: High dose radiotherapy; Standard radiotherapy
Radiation: 2.15 gray and 1.8 gray. Max. 5 weeks.
  Arms: Low dose radiotherapy

SUMMARY:
The purpose of this study is to maximize patient involvement in the treatment of anal cancer. Specifically, the investigators will investigate whether patients wish to take part in the decision making on radiation dose and whether they want a high or low radiation dose.

DETAILED DESCRIPTION:
The study will also provide new knowledge on the effect and side effects of irradiation of anal cancer, and detailed data from the dose planning will be instrumental in optimizing future decision aids.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma of the anal duct or perianal (non-hairy skin, max 5 cm from the anal verge)
* T2-T4 N0-3
* Age ≥ 18 years
* Performance status 0-2
* Sufficient organ and bone marrow function defined as:

  * Neutrophils ≥ 1.5 x 10^9/L
  * Thrombocytes ≥ 100 x 10^9/L
* Curative intent radiation treatment deemed possible
* Patients chooses 1 of 3 options:

  * I do not wish to decide on details of my treatment, but I would like to receive the standard treatment
  * I want to receive the high radiation dose
  * I want to receive the low radiation dose
* Written and orally informed consent

Exclusion Criteria:

* Non-resectable metastases
* Tumor > 10 cm or the total tumor volume (incl. lymph node metastases) is too large to be included in an appropriate radiation field (after possible neoadjuvant chemotherapy)
* Pregnant or breastfeeding women
* Fertile women not willing to use effective contraception
* Serious co-morbidity that would hinder interfere with radiation treatment or hinder patient compliance (e.g. incapacity to understand or complete questionnaires)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2025-06 (Actual)

PRIMARY OUTCOMES:
The fraction of enrolled patients wanting to take part in the decision making on radiation dose level | 6 months after the last patient has finished radiotherapy
The fraction of enrolled patients choosing the lower radiation dose | 6 months after the last patient has finished radiotherapy

SECONDARY OUTCOMES:
Number of patients with a V45Gy of less than 300 cc for the small bowel calculated on the basis of dose plans | 6 months after the last patient has finished radiotherapy
Number of patients with a V35Gy of less than 75% for the bladder calculated on the basis of dose plans | 6 months after the last patient has finished radiotherapy
Number of patients with treatment related adverse events as assessed by healthcare staff based on the common toxicity criteria (CTCAE v.4.0) | 5 years after inclusion of the last patient
Quality of life as assessed by combined questionnaires EORTC QLQ CR30 and CR29 | 5 years after inclusion of the last patient
Subjective symptoms as assessed by LARS score (low anterior resection syndrome) | 5 years after inclusion of the last patient
Rate of complete response | 6 months after the last patient has finished radiotherapy
Number of patients with loco-regional recurrence 60 months after end of treatment | 5 years after inclusion of the last patient
Number of patients with distant metastases at 5 years | 5 years after inclusion of the last patient
Colostomy free survival | 5 years after inclusion of the last patient
Disease free survival | 5 years after inclusion of the last patient
Overall survival | 5 years after inclusion of the last patient
Number of patients with HPV at time of enrollment | 6 months after the last patient has finished radiotherapy
Response evaluation assessed by diffusion weighted imaging | 6 months after the last patient has finished radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Lars H Jensen, MD,PhD, Study Chair — Vejle Hospital
Locations (1):
- Vejle Hospital, Vejle, Denmark